CLINICAL TRIAL: NCT04352400
Title: RAndomized Clinical Trial in COvid19 Patients to Assess the Efficacy of the Transmembrane Protease Serine 2 (TMPRSS2) Inhibitor NAfamostat (RACONA Study)
Brief Title: Efficacy of Nafamostat in Covid-19 Patients (RACONA Study)
Acronym: RACONA
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Padova (Other)
Collaborators: Yokohama City University (Other); University of Zurich (Other)
Responsible Party: Principal Investigator, Gian Paolo Rossi, MD, FAHA, FACC, Prof., University Hospital Padova
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RACONA Nafamostat
Record Dates: First submitted 2020-04-03; First posted 2020-04-20 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: COVID19
Keywords: Nafamostat; proteases; TMPRSS2; covid-19; coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — nafamostat

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, placebo-controlled parallel-group trial, on top of best standard of care
Who Masked: Participant, Investigator
Masking Description: Randomization will be done with an algorithm tailored to the study design. Investigators and patients will be blinded to the treatment administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nafamostat (Active Comparator): Nafamostat mesylate on top of best standard of care.
  Interventions: Drug: Nafamostat Mesilate
- Placebo (Placebo Comparator): Placebo on top of best standard of care.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nafamostat Mesilate — administered intravenously as a continuous infusion
  Other Names: no alternative name. Commercial brands are available.
  Arms: Nafamostat
Drug: Placebo — administered intravenously as a continuous infusion
  Other Names: no alternative name.
  Arms: Placebo

SUMMARY:
RACONA is a prospective trial that will test the hypothesis that nafamostat can lower lung function deterioration and need for intensive care admission in COVID-19 patients.

Design: Adult hospitalized COVID-19 patients will be randomized in a prospective double-blind randomized placebo-controlled study to test the clinical efficacy of nafamostat mesylate (administered intravenously) on top of best standard of care.

Primary outcome measures: the time-to-clinical improvement, defined as the time from randomization to an improvement of two points (from the status at randomization) on a seven category ordinal scale or live discharge from the hospital, whichever comes first.

DETAILED DESCRIPTION:
Purpose: SARS-Cov-2 enters the lung cells by binding to ACE-2 and activating the protease TMPRSS2, which, therefore, can be a target for antiviral treatment. Accordingly, TMPRSS2 inhibitors prevent SARS-CoV cell entry in vitro. The most potent such inhibitors, nafamostat is being used as anticoagulant and anti-pancreatitis agent, and is approved for the treatment of cystic fibrosis as its mucolytic action can prevent lung function deterioration by owering airways infections.

RACONA study will test the hypothesize that nafamostat is useful in COVID-19 lung involvement because COVID-19 entails activation of the coagulation cascade, pulmonary embolism, and bacterial superinfections.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized, COVID-19 positive, between 18 and ≤ 85 years of age;
* Signed Inform Consent Form;
* Body temperature > 37.3 ℃;
* Oxygenation criterion (any of the following): i) Oxygen saturation ≤94% on Room Air; ii) PaO2/FiO2 ratio ≤300 mmHg but > 100 mmHg, if patient on supplemental oxygen; iii) SpO2/FiO2<200 if no arterial blood gas available;
* Respiratory rate (RR) ≥ 25 beats/min.

Exclusion Criteria:

* Pregnant or lactating females;
* Unwillingness or inability to complete the study.
* Rapidly deteriorating clinical condition or low likelihood to complete the study according to the investigator;
* eGFR < 30 ml/min/m2 assessed with CKD EPI formula;
* Current or chronic history of liver disease (Child Pugh score ≥ 10), or known hepatic or biliary abnormalities;
* Participation in a clinical trial with an investigational product within the following time period prior to the first dosing day in the current study: 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer);
* Patients requiring high doses of loop diuretics (i.e. > 240 mg furosemide daily) with significant intravascular volume depletion, as assessed clinically;
* History of allergy;
* History of sensitivity to heparin or heparin-induced thrombocytopenia;
* Unstable hemodynamics in the preceding 4 hours (SBP < 90 mmHg, and/or vasoactive agents required);
* Hemoglobin < 7 at time of drug infusion. Transfusion is allowed to increase hemoglobin levels before entry into the study;
* Malignancy or any other condition for which estimated 6-month mortality >50%;
* Arterial blood pH less than 7.2;
* Known evidence of chronic interstitial infiltration at imaging;
* Known hospitalization within the past six months for respiratory failure (PaCO2 > 50 mmHg or PaO2 < 55 mmHg, or oxygen saturation <88% on FiO2 = 0.21);
* Known chronic vascular disease resulting in severe exercise restriction (i.e. unable to perform household duties);
* Known secondary polycythemia, severe pulmonary hypertension, or ventilator dependency;
* Known vasculitis with diffuse alveolar hemorrhage;.
* Pre-existing renal failure on hemodialysis or peritoneal dialysis requiring renal replacement therapy;
* Extracorporeal membrane oxygenation (ECMO);
* Immunosuppressive treatment;
* Patient in trials for COVID-19 within 30 days before;
* Unstable hemodynamics in the preceding 4 hours (MAP ≤ 65 mmHg, or SAP < 90 mmHg, DAP < 60 mmHg, and vasoactive agents required);
* Hyperkalemia , i.e. serum K+ levels > 5.0 mEq/L;
* Severe active bleeding;
* Any other uncontrolled comorbidities that increase the risks associated with the study drug administration, as assessed by the medical expert team.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2021-06-04 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Time-to-clinical improvement | day 1 until day 28
  Time-to-clinical improvement (time from randomization to an improvement of two points (from the status at randomization) on a 7 category ordinal scale or live discharge from the hospital, whichever came first.

SECONDARY OUTCOMES:
Responders | day 1 until day 28
  Rate of patients showing improvement of 2 points in 7 category ordinal scale (with 7 points the worst)(PubMed ID: 32187464)
Critical or dead patients | day 1 until day 28
  Proportion of patients who will progress to critical illness/death
pO2/FiO2 ratio | day 1 until day 28
  Change in pO2/FiO2 ratio over time
SOFA score over time | day 1 until day 28
  Change Sequential organ failure assessment score (SOFA score) over time. The Score ranges from 0 to 24 (with 24 the worst)(PubMed ID: 11594901)
Hospitalization | day 1 until day 28
  Duration of hospitalization in survivors (days)
Mechanical ventilation | day 1 until day 28
  Number of patients who require ventilation
Mechanical ventilation duration | day 1 until day 28
  Duration of ventilation (days)
Cardiovascular disease | day 1 until day 28
  Proportion of patients who develop arrhythmia, or myocardial infarction, or other cardiovascular disease not present at the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Gian Paolo Rossi, Prof., Principal Investigator — University of Padova, Italy
Locations (1):
- Azienda Ospedale Università di Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yamamoto M, Matsuyama S, Li X, Takeda M, Kawaguchi Y, Inoue JI, Matsuda Z. Identification of Nafamostat as a Potent Inhibitor of Middle East Respiratory Syndrome Coronavirus S Protein-Mediated Membrane Fusion Using the Split-Protein-Based Cell-Cell Fusion Assay. Antimicrob Agents Chemother. 2016 Oct 21;60(11):6532-6539. doi: 10.1128/AAC.01043-16. Print 2016 Nov. PMID 27550352
- [Result] Hoffmann M, Kleine-Weber H, Schroeder S, Kruger N, Herrler T, Erichsen S, Schiergens TS, Herrler G, Wu NH, Nitsche A, Muller MA, Drosten C, Pohlmann S. SARS-CoV-2 Cell Entry Depends on ACE2 and TMPRSS2 and Is Blocked by a Clinically Proven Protease Inhibitor. Cell. 2020 Apr 16;181(2):271-280.e8. doi: 10.1016/j.cell.2020.02.052. Epub 2020 Mar 5. PMID 32142651
- [Result] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Result] Cao B, Wang Y, Wen D, Liu W, Wang J, Fan G, Ruan L, Song B, Cai Y, Wei M, Li X, Xia J, Chen N, Xiang J, Yu T, Bai T, Xie X, Zhang L, Li C, Yuan Y, Chen H, Li H, Huang H, Tu S, Gong F, Liu Y, Wei Y, Dong C, Zhou F, Gu X, Xu J, Liu Z, Zhang Y, Li H, Shang L, Wang K, Li K, Zhou X, Dong X, Qu Z, Lu S, Hu X, Ruan S, Luo S, Wu J, Peng L, Cheng F, Pan L, Zou J, Jia C, Wang J, Liu X, Wang S, Wu X, Ge Q, He J, Zhan H, Qiu F, Guo L, Huang C, Jaki T, Hayden FG, Horby PW, Zhang D, Wang C. A Trial of Lopinavir-Ritonavir in Adults Hospitalized with Severe Covid-19. N Engl J Med. 2020 May 7;382(19):1787-1799. doi: 10.1056/NEJMoa2001282. Epub 2020 Mar 18. PMID 32187464
- [Result] Minakata D, Fujiwara SI, Ikeda T, Kawaguchi SI, Toda Y, Ito S, Ochi SI, Nagayama T, Mashima K, Umino K, Nakano H, Yamasaki R, Morita K, Kawasaki Y, Sugimoto M, Yamamoto C, Ashizawa M, Hatano K, Sato K, Oh I, Ohmine K, Muroi K, Ohmori T, Kanda Y. Comparison of gabexate mesilate and nafamostat mesilate for disseminated intravascular coagulation associated with hematological malignancies. Int J Hematol. 2019 Feb;109(2):141-146. doi: 10.1007/s12185-018-02567-w. Epub 2018 Dec 8. PMID 30536180
- [Result] Yu G, Li S, Wan R, Wang X, Hu G. Nafamostat mesilate for prevention of post-ERCP pancreatitis: a meta-analysis of prospective, randomized, controlled trials. Pancreas. 2015 May;44(4):561-9. doi: 10.1097/MPA.0000000000000310. PMID 25822153
- [Result] Ferreira FL, Bota DP, Bross A, Melot C, Vincent JL. Serial evaluation of the SOFA score to predict outcome in critically ill patients. JAMA. 2001 Oct 10;286(14):1754-8. doi: 10.1001/jama.286.14.1754. PMID 11594901
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208
- [Derived] Flumignan RL, Tinoco JDS, Pascoal PI, Areias LL, Cossi MS, Fernandes MI, Costa IK, Souza L, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Prophylactic anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD013739. doi: 10.1002/14651858.CD013739. PMID 33502773
- Available data/document: Individual Participant Data Set: GPR (PI) — https://ncov.medsci.ox.ac.uk — The link https://ncov.medsci.ox.ac.uk allows connection to EDCap database, a secure web platform for building and managing online databases and surveys. Data collection will use the WHO Case Record Form.